Low-Carbohydrate Diabetes Prevention Program Among Veterans With Prediabestes (VA LC-DPP)

Prepared for ClinicalTrials Resubmission 4/20/21

### Statistical Analysis Plan:

### Quantitative analysis

Descriptive statistics will be used for baseline survey response data including demographic and socioeconomic characteristics. For all continuous outcomes, we will calculate mean change and standard deviation from baseline to 6 months and 12 months and compare outcomes from baseline to 6 months and 12 months using paired t-tests. For all categorical outcomes, we will IRB Protocol Template – VAAAHS\_021419 Page 14 of 18 use chi-square or Fisher's exact tests to examine changes from baseline to 6 and 12 months. All analyses will be conducted using Stata 14.

### Qualitative analysis:

Semi-structured interviews will be recorded and transcribed verbatim. Interviews will then be imported into qualitative analysis software. Two investigators will independently read and code transcribed interviews. Interviews will then be coded jointly using consensus conferences. Interviews will be analyzed using directed content analysis 27, which is to say that codes will be created to reflect the main topics in the interview guide and to characterize the patterns and themes that emerged from the data.28

# Cravings: Control of Eating Questionnaire

#### Over the past 7 days...

How Q1 Answer Items on Dalton M, strong choices the CoEQ Finlayson on a G, Hill A, was your are desire to sliding assessed Blundell J. eat sweet scale by 100 Preliminar

foods? from 0 to mm VAS y

100 with with validation

anchors items and at 0 and relating to principal

100: each compone

How Q2 0- not at subscale nts strong all strong being analysis was your 10 averaged of the desire for 20 to create Control of

Over the past 7 days, how often have you had cravings f

Sweet Q3 Answer foods like choices Other on a Q4 sliding sweet scale foods from 0 to (cakes, 100 with pastries, anchors cookies, etc)? at 0 and 100: Fruit or Q5 0- not at fruit all juice?

non-

Dairy Q6 10 foods 20 (cheese, 30 yogurts, 40 milk, etc)?

60

 Starchy
 Q7
 70

 Foods
 Q8
 80

 that are
 90

 not sweet
 100

like extremely often

French fries, potato chips,

**Stress Eating** 

#### Please indicate how you usually experience a stressful ev

| I eat more Q1 | Answer | Reverse | Tsenkova, |
|---------------|-----------|-----------|------------|
| of my | choices 1 | code and | V., |
| favorite | through 4 | sum, so | Boylan, J. |
| foods to | with | that | M., & |
| l eat more Q2 | anchors | higher | Ryff, C. |
| than I | on 1 and | scores | (2013). |
| ucually | 4: | indicated | Stress |

Below is a list of reasons that people sometimes give for eating tasty foods and drinks such as:

- Sweets like chocolate, doughnuts, cookies, cake, candy, ice cream, other desserts.
- Salty snacks like chips, pretzels, and crackers.
- Fast foods like hamburgers, cheeseburgers, pizza, fried chicken and French fries.
- Sugary drinks like soda, sweet tea, milkshakes, and

| To forget y Q3 | 1 = | Coping | Burgess, |
|----------------|----------|-----------|------------|
| Because it Q4 | Almost | score: | E. E., |
| To cheer u Q5 | never/Ne | Average | Turan, B., |
| To forget a Q6 | ver | of four | Lokken, K. |
| | 2 = Some | responses | L., Morse, |
| | of the | | Δ & |

## **Energy Levels between Meals**

#### In the past week, two hours after you ate BREAKFAST, h

| Alert | Q1 | Answer | NA | NA |
|-------------|------|-----------|----|----|
| Energetic | Q2 | choices 1 | | |
| Tired | Q3 | through | | |
| Brain fog o | Q4 | 7, with | | |
| Food cravi | ıQ5 | anchors | | |
| Hunger | Q6 | on 1, 7: | | |
| Moodines | s Q7 | 1- Not at | | |
| | | all | | |
| | | 2 | | |

## In the past week, two hours after you ate LUNCH, how n

NA

| Alert | Q8 | Answer |
|-------------|-------|-----------|
| Energetic | Q9 | choices 1 |
| Tired | Q10 | through |
| Brain fod o | Q11 | 7, with |
| Food cravi | ıQ12 | anchors |
| Hunger | Q13 | on 1, 7: |
| Moodines | s Q14 | 1- Not at |

#### **Physical Symptoms**

How often have you experienced the following over the

Acne Q1 NA NA

Bad breath Q2 Bloating or Q3 Cold hands Q4
Constipatic Q5
Diarrhea Q6
Dizziness Q7
Dry mouth Q8
Constant tl Q9
Food pain (Q10

#### Headaches Q11

Heart Q12
palpitatio
ns or a
racing
heart
Heartburn Q13
Joint or Q14
muscle
pain
Muscle Q15

cramps Not at all Nausea Q16 1 day a Trouble Q17 week concentra 2-3 days ting a week Weakness Q18 4-5 days a week

Hair loss Q19 6-7 days a
Sexual Q20 week
problems
Numbnes Q21
s (loss of

in the
feet, legs,
or hands
Tingling Q22
or
prickling
sensation
s in the
feet, legs,
or hands

sensation)

Burning Q23

or

shooting

pain in

the feet,

legs, or

hands

Blurred or Q24

deteriorat

ing vision

Please Q25 describe any other psycholog ical or physical

Participa nts may enter free text of whatever they

choose.

symptom s that you experienc ed during the past

month.

# Health Global Health PROMIS Questionnaire:

## Please respond to each item by marking one box per rol

| | | | g <u>5</u> | , ,, , |
|---|---|---|---|---|
| In | Q1 | 5- | Re-code: | PROMIS |
| In | Q2 | Excellent | Q7 (pain | Health |
| general, | | 4- Very | on | Organizati |
| would | | good | average): | on and |
| you say | | 3- Good | 0 = 5 | PROMIS |
| your | | 2- Fair | 1,2,3 = 4 | Cooperati |
| quality of | | 1- Poor | 4,5,6 = 3 | ve Group, |
| life is: | | | 7,8,9 = 2 | 2008- |
| In | Q3 | | 10 = 1 | 2012. |
| general, | | | | https://w |
| how | | | Global | ww.iconq |
| would | | | Physical | uerms.org |
| you rate | | | Health | /sites/all/ |
| your | | | Score: | files/attac |
| physical | | | Sum | hments/p |
| health? | | | responses | dfs/PROM |
| In | Q4 | | to 3, 6, 7, | ISGlobalH |
| general, | | | 8. | ealthScale |
| how | | | Fatigue | V1.0- |
| would | | | on | 1.1.pdf |
| you rate | | | average, | |
| your | | | pain on | |
| mental | | | average, | |
| health, | | | extent to | |
| including | | | carry out | |
| your | | | physical | |

activities, how

would

you rat

mood and

ability to

think?

your

In Q5 eyour general, physical how health.

Global you rate Mental your Health satisfactio score: n with SUM: 2, 4, your social 5, 10 How activities often and bothered relationsh by ips?

emotional Q6 In problems, general, rate your please mental rate how health, well you rate your carry out satisfactio your usual n, quality social of life.

acivities and roles. (This includes activities at home, at work and in your communit y, and responsibi lities as a parent, child, spouse, employee , friend,

etc.)

To what Q7 5-

extent are Completel

you able y

to carry 4- Mostly

out your 3-

everyday Moderate

physical ly

activities 2- A little such as 1- Not at walking, all

climbing stairs, carrying groceries, or moving a chair?

## *In the past 7 days:*

How Q8 5- Never often 4- Rarely

have you 3-

been Sometime

bothered s

by 2- Often emotional 1- Always

problems such as feeling anxious, depressed

, or irritable?

How Q9 5- None would 4- Mild you rate 3-

your Moderate fatigue on 2- Severe average? 1- Very severe

How Q10 Answer would choices 0 through you rate your pain 10 with on anchors average? on 0, 10: 0- No pain 1 2 3 4 5 6 7 8 9 10- Worst pain

#### **Program Evaluation** How Q1 Answer NA NA would choices 1-7 with you rate your anchors overall on 1,7: satisfactio 1- Not at n with the all program? satisfied 2 3 4 5 6 7- Very satisfied If a friend Q2 1- No, were in definitely need of not similar 2- No, not

imaginabl

e

What's Q3
the most
meaningf
ul thing
you've
learned or
gotten
out of this
program?

Q4

Participa nts may enter free text of whatever they choose.

How helpful have the classes been?

Answer choices 1-7 with anchors on1,7:

1- don't include them, they were not helpful

ne 2

3

4

5

6

7- you must include them, they were very helpful Do you Q5

have any
suggestio
ns about
how we
can
improve
the

the classes? Which were your favorite or least favorite topics?

How Q6 Answer helpful choices 1were the 7 with handouts anchors ? How 1,7: 1- don't much would include you them, they were recomme nd that not we helpful include 2 them in 3 4 the next study? 5 6 7- you

> must include them, they were very helpful

Do you Q7 Participa have any nts may suggestio enter free ns about text of how we whatever can they improve choose.

the

handouts? Which were your favorite or least favorite topics?

## **Social Support**

## How often in the last 30 days has your family or friends

| Q1 | 1 = | Average | Norman, |
|---|---|---|---|
| Q2 | Almost | responses | G. J., |
| Q3 | never | of the 6 | Carlson, J. |
| | 2 = Once | questions. | A., Sallis, |
| | in a while | **NOTE: | J. F., |
| | 3 = | this just | Wagner, |
| | Sometime | appears | N., Calfas, |
| Q4 | S | to be how | K. J., & |
| | 4 = Often | it is in the | Patrick, K. |
| | 5 = | scoring, | (2010). |
| | Almost | but | Reliability |
| Q5 | always | doesn't | and |
| | | actually | validity of |
| | | say how | brief |
| | | to do it. | psychosoc |
| Q6 | | | ial |
| | | | measures |
| | | | related to |
| | | | dietary |
| | | | behaviors. |
| | Q2<br>Q3<br>Q4 | Q2 Almost Q3 never 2 = Once in a while 3 = Sometime Q4 s 4 = Often 5 = Almost Q5 always | Q2 Almost responses Q3 never of the 6 2 = Once questions. in a while **NOTE: 3 = this just Sometime appears Q4 s to be how 4 = Often it is in the 5 = scoring, Almost but Q5 always doesn't actually say how to do it. |

## **Open Ended Support**

Have you Q1 Participa NA NA

gotten nts may
any enter free
feedback text of
from whatever
family, they
friends, or choose.

physicians /healthcar

e

providers about this program or your experienc e with it? If so, what did

they say?

## **Medication Changes**

# 6- month question

Did any of Q1 Yes/No

your

medicatio

ns or doses change since starting

starting this

program?

If yes, Free text

please specify which medicatio

ns were changed or added.

If yes, Q2 Increased
was the Decrease
dose d
increased I don't
or know
decreased
?

12month question

Did any of Q1 Yes/No your medicatio ns or doses change over the past 6 months program (i.e. maintena nce phase)? If yes, Free text please specify which medicatio ns were changed or added. If yes, Q2 Increased was the Decrease dose d I don't increased or know decreased ?

How Q1 Answer NA NA much do choices 1-

| How much do you think this diet has improved your physical health? How much do you think this diet has | Q2<br>Q3 | 7 with anchors 1,7: 1- Not at all 2 3 4 5 6 7- Very much so |
|---|---|---|
| How hard<br>is it to<br>stay on<br>your diet? | Q4 | Answer choices 1-7 with anchors 1,7: 1- Very easy 2 |
| How<br>often do<br>you cheat<br>on your<br>diet? | Q5 | Answer choices 1- 7 with anchors 1,7: 1- Not at all 2 3 4 5 6 7- Very often Open Ended Diet |

When you Q1 Participa NA NA

follow nts may
this low- enter free
carbohydr text of
ate food whatever
plan: they
What choose.

about your health got better?

When you Q2 Participa follow nts may this low-carbohydr text of ate food whatever plan: they What choose.

about your health got worse? When you Q3a Answer follow options 1-this low- 7 with carbohydr anchors ate food given at plan, how 1,4,7: much do

you tend 1- Much to pay for less food? money than

before 2 3

4- About the same as before

5 6

7- Much more money than before

Why or Q3b why not?

Participa nts may enter free text of whatever they choose.

## **Treatment Self-Regulation Questionnaire**

## There are a variety of reasons why patients may take

Because I Q1 Answer Autonom Williams feel that I options 1- ous score: et al. want to 7 with Average Healthanchors responses Care, Selftake responsibi given at for items Determin lity for my 1,4,7: 1, 3, 6, 8, ation own 11, 13. Theory health. 1- Not Questionn Because I Q2 true at all Controlle aire

would 2 d score: Packet via feel guilty 3 Average selfdeter or 4responses minationt Somewha for items: heory.org ashamed

of myself t true 2, 4, 7, 9, if I didn't 5 12, 14.

take steps 6

7- Very to Amotivati prevent true on score: diabetes. Average Because I Q3 responses personally for items believe it 5, 10, 15.

is the best thing for my health.

Because Q4

others would be upset with me if I didn't take steps

to

prevent diabetes.

Q5 I really

don't think about it.

Because I Q6

have carefully thought about it and is very

believe it

important for many

aspects of

my life.

Because I Q7

would

feel bad

about

myself if I

didn't

take steps

to

prevent

diabetes

Because it Q8

is an

important

choice I

really

want to

make.

Because I Q9

feel

pressure

from

others to

take steps

to

prevent

diabetes

Because it Q10

is easier

to do

what I am

told than

think

about it.

## Because it Q11

is

consistent

with my

life goals.

Because I Q12

want

others to

approve

of me.

Because it Q13

is very

important

for being

as healthy

as

possible.

Because I Q14

want

others to

see I can

do it.

I don't Q15

really

know

why.

### **Physical Activity Questionnaire**

#### Think about all the vigorous activities which take hard

During Q1 *Participa* Scored by Craig et the last 7 *nts may* taking the al.

days, on *enter* sum of Internatio

how days per time nal many week (hours Physical days did including: and Activity 0-7 you do minutes) Questionn vigorous 8: Don't and then aire: 12physical Know/Not weighting Country activities? Sure values Reliability

9: according and

Refused to Validity.

activity

average 2003.

How Q2 *Participa* MET much *nts enter* values for

time did values in vigorous, you two moderate usually boxes: and

spend Hours per walking. doing day: Weighted vigorous Minutes values physical per day: summed activities to get on one of final those physical

Now think about activities which take moderate

During Q3 Participan the last 7 ts may days, on enter how days per many week days did including: you do 0-7 moderate 8: Don't

days?

physical

activities? Sure

9:

Refused

Know/Not

Q4 Participa How much nts enter time did values in you two usually boxes: spend Hours per doing day: moderate Minutes physical per day:

activities on one of those days?

## Now think about the time you spent walking in the last

Q5 During Participan the last 7 ts may days, on enter how days per many week days did including: 0-7 you walk for at 8: Don't Know/Not least 10 minutes Sure 9: at a time.

Refused

How Q6 Participa much nts enter time did values in you two usually boxes: spend Hours per walking day: on one of Minutes those per day:

days?

Now think about the time you spent sitting on week

Participa During Q7 the last 7 nts enter values in days, how much two time did boxes: you Hours per usually day: spend Minutes sitting on per day:

a week day?

## **Fatigue**

#### During the past 7 days...

I feel 1 = Not at Sum Kemper-Q1 fatigued responses Gascon, I have Q2 2 = A little of the Global four Health trouble bit questions and Wellstarting 3 = Somewha for the being. The things because I raw score. Ohio am tired 4 = Quite Included State In the past 7 days... a bit on PDF is University 5 = Very How run Q3 the . (See down did much conversio PDF) you feel n chart to on determin average? e the T-Q4 How score.

## **Sleep Disturbance**

#### In the

| My sleep<br>quality | Q1 | 5 = Very<br>poor | Sum responses | Kemper-<br>Gascon, |
|---|---|---|---|---|
| was | | 4 = Poor | of the | Global |
| | | 3 = Fair | four | Health |
| | | 2 = Good | questions | and Well- |
| | | 1 = Verv | for the | being. The |
| In the | | | raw score. | Ohio |
| My sleep | Q2 | 5 = Not at | Included | State |
| was | | all | on PDF is | University |
| refreshing | | 4 = A little | the | . (See |
| | | bit | conversio | PDF) |
| | | 3 = | n chart to | |
| I had a | Q3 | 1 = Not at | determin | |

I had Q4 all e the Tdifficulty 2 = A little score.

falling bit asleep 3 =

## **Demographics**

NA

Do you Q1
have any
significant
medical
diagnosis,
surgery,
hospitaliz

Participa NA
nts may
enter free
text of
whatever
they
choose.

ations, or other major health issue? If so, please describe. Do you Q2 Participa take nts may metformi enter free n for your text of diabetes? whatever (It's also they called choose.

Glucopha

ge,

Glumetza,

and

Fortamet. If so, how

much

(total) do

you take

per day?

For

example,

you might

take 500

or

2,000mg

a day.

What Q3 Participa other nts may Over the Q4 Participa past 7 nts may days, how enter free many text of cigarettes whatever have you they smoked choose.

per day on

average?

What is Q5 Some the high highest school level of High formal school education graduate you have Some complete college d? College

graduate
Some
postcollege
education
Master's
degree
PhD
degree

What is Q6 Single, How long Q7 Sliding have you scale had type from 0-50 2 years diabetes, with in years? anchors every 5 years.

What is yo Q8 Text box w How old ar Q9 18-25 26-35

What is yo Q10 Participant What is yo Q11 Participant

What is yo Q12 Male
Are you Hi: Q13 Yes
No

What is Q14 White
your race Black or
or ethnic African
backgrou American
nd? Check American
ALL that Indian or
apply. Alaska

Native
Asian
Native
Hawaiian
or Pacific
Islander
Other
Prefer not
to answer

8th grade

## What is the Q15

or less Some high school but did not graduate High school graduate or GED Some college or a 2-year degree 4-year college graduate More than 4year college degree Prefer not

to answer

| What is | Q16 | Less than |
|----------|-----|-----------|
| your | | \$10,000 |
| annual | | \$10,000- |
| total | | \$19,999 |
| househol | | \$20,000- |
| d income | | \$29,999 |
| from all | | \$30,000- |
| sources | | \$39,999 |
| before | | \$40,000- |
| taxes? | | \$49,999 |
| | | \$50,000- |
| | | \$59,999 |
| | | \$60,000- |
| | | ¢60 000 |

Treatment Self-Regulation
Questionnaire
There are a variety of reasons why
patients may take steps to prevent
diabetes. Please consider the
following behaviors and indicate
how true each of these reasons is
for you. The reason I would take
steps to prevent diabetes is:

Because I feel that I want to take responsibility for my own health. Q1 Because I would feel guilty or ashamed of myself if I didn't take steps to prevent diabetes. Q2 Because I personally believe it is the best thing for my health. Q3 Because others would be upset with me if I didn't take steps to prevent diabetes. Q4 I really don't think about it. Q5

Answer options 1- Autonomous 7 with score: anchors Average given at responses for 1,4,7: items 1, 3, 6, 8, 11, 13. Williams 1- Not et al. true at all Controlled score: Health-2 Care, Self-Average 3 responses for Determin 4items: 2, 4, 7, 9, ation Somewha 12, 14. Theory t true Questionn 5 Amotivation aire 6 Packet via score: 7- Very Average selfdeter responses for true minationt items 5, 10, 15. heory.org

| Because I have carefully thought about it and believe it is very | |
|------------------------------------------------------------------|-----|
| important for many aspects of my | |
| life. | Q6 |
| Because I would feel bad about myself if I didn't take steps to | |
| prevent diabetes | Q7 |
| Because it is an important choice I | |
| really want to make. | Q8 |
| Because I feel pressure from others | |
| to take steps to prevent diabetes | Q9 |
| Because it is easier to do what I am | |
| told than think about it. | Q10 |
| Because it is consistent with my life | 011 |
| goals. Because I want others to approve of | Q11 |
| me. | Q12 |
| Because it is very important for | |
| being as healthy as possible. | Q13 |
| Because I want others to see I can | |
| do it. | Q14 |
| I don't really know why. | Q15 |